CLINICAL TRIAL: NCT02838992
Title: Multi-center Clinical Study of Immunosuppressants, Cyclophosphamide, And Cord Blood Transfusion in Treating Patients With Severe Aplastic Anemia
Brief Title: ATG Combined With Cyclophosphamide And Cord Blood Transfusion in Treating Patients With Severe Aplastic Anemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinan Military General Hospital (Other)
Collaborators: Shandong University of Traditional Chinese Medicine (Other); Jining Medical University (Other); Weifang Medical University (Other); Guangzhou First People's Hospital (Other); Harbin Hematology and Oncology Institute (Other); Jining First People's Hospital (Other); JIANGXI Provincal People's Hospital (Unknown); Jinhua Central Hospital (Other); Linyi People's Hospital (Other); Shandong Cord Blood Bank (Unknown); Qingdao Hiser Medical Group (Other); Qingdao University (Other); Taian City Central Hospital (Other); Yantai Yuhuangding Hospital (Other); Yishui Central Hospital of LINYI (Unknown); Institute of Hematology & Blood Diseases Hospital, China (Other); Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Fang Zhou, Principal Investigator, Jinan Military General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JinanMGH
Record Dates: First submitted 2016-07-06; First posted 2016-07-20 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Aplastic Anemia
Keywords: Cyclophosphamide; Umbilical Cord Blood; ATG
MeSH Terms: conditions — Anemia, Aplastic | interventions — thymoglobulin; Antilymphocyte Serum; Cyclophosphamide; Cyclosporins; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG, Cy and cord blood transfusion group (Experimental): ATG 3mg/kg/d for 5 days Cy 50mg/kg/d for 2 days CSA Started from 5mg/kg/d and adjusted to maintain trough serum concentration of 200-400ng/ml One unit of cord blood having no more than 3 HLA-A,B and DRB1 mismatches is transfused 24h after last dose of ATG administration.
  Intervention:
  Drug: Rabbit ATG, Thymoglobuline (Genzyme) plus Cyclophosphamide plus CSA Biological: Cord blood transfusion
  Interventions: Drug: Rabbit ATG, (Genzyme); Drug: Cy; Drug: CsA; Biological: Cord blood
- ATG and CSA group (Active Comparator): ATG 3mg/kg/d for 5 days CSA started from 5mg/kg/d and adjusted to maintain trough serum concentration of 200-400ng/ml Intervention: Drug: Rabbit ATG, Thymoglobuline (Genzyme) plus CSA
  Interventions: Drug: Rabbit ATG, (Genzyme); Drug: CsA

INTERVENTIONS:
Drug: Rabbit ATG, (Genzyme) — ATG is an infusion of rabbit-derived antibodies against human T cells, which is used in the prevention and treatment of acute rejection in organ transplantation and therapy of aplastic anemia
  Other Names: Thymoglobuline; Anti-thymoeyteGlobulin
Drug: Cy — Cyclophosphamide is a medication mainly used in chemotherapy. It is an alkylating agent of the nitrogen mustard type
  Other Names: Cyclophosphamide; Cytophosphane
  Arms: ATG, Cy and cord blood transfusion group
Drug: CsA — CsA is an immunosuppressant drug widely used in organ transplantation to prevent rejection. It reduces the activity of the immune system by interfering with the activity and growth of T cells
  Other Names: Ciclosporin A; Cyclosporine
Biological: Cord blood — Cord blood is blood that remains in the placenta and in the attached umbilical cord after childbirth. Cord blood is collected because it contains stem cells, which can be used to treat hematopoietic and genetic disorders
  Other Names: Umbilical cord blood
  Arms: ATG, Cy and cord blood transfusion group

SUMMARY:
To assess whether ATG Combined With Cyclophosphamide and cord blood infusion can accelerate hematopoietic reconstruction in severe aplastic anemia patients and improve clinical curative effect and safety

DETAILED DESCRIPTION:
Aplastic Anemia( AA), is a set of bone marrow hematopoietic dysfunction caused by a variety of causes, with hyperplasia of bone marrow hematopoietic cells to reduce whole blood cells and peripheral blood at the characteristics of clinical main performance for anemia, bleeding and infection. According to the severity of the bone marrow failure and the progress of the clinical course ,it is divided into Severe Aplastic Anemia (SAA) and the Non - Severe Aplastic Anemia (NSAA).Severe Aplastic Anemia can be divided into two categories: Very Severe Aplastic Anemia (VSAA) and Severe Aplastic Anemia (SAA), with the characteristics of rapid progress, refractory, poor prognosis, high mortality .The natural course is six months or so, and most patients die in a year . Hematopoietic stem cell transplantation and immunosuppressive therapy are two main treatment . The former is by far the only possible cure. It is recommended as first-line treatments, if patients have a matched sibling donor. The recommended age limit is 40 years old. But for those who have no sibling donor or patients older than 40 years old, it is recommend the immunosuppressive therapy.

The investigators have already summarized the effectiveness of rabbit antithymocyte immunoglobulin (ATG), cyclophosphamide (Cy) and cyclosporine, A (CsA) and the combination of the umbilical cord blood infusion for SAA/VSAA patients without suitable donor, with short duration, without long-term immunosuppressive therapy history. The total effectiveness rates has improved to 88%, with shorter immunosuppressive maintaining therapy , rapid hematopoietic reconstruction, fewer complications. The aim of this study is to further explore whether this solution can accelerate hematopoietic reconstruction of SAA/VSAA patients and its clinical curative effect and security. This study scheme has been approved by the Jinan military region general hospital medical ethics committee.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ,under the age of 60.
2. Diagnosis of SAA and VSAA in accordance with the <aplastic anemia, diagnosis and treatment expert consensus> Camitta standard (see appendix 1).
3. Confirmed of heavy and very heavy aplastic anemia within 6 months.
4. No obvious abnormal liver and kidney function: ALT, AST,≤2.5 times the upper limit of normal , serum Creatinine and BUN ≤1.25 times the upper limit of normal
5. Clear understanding, voluntary to participate in the study, and signed informed consent document by the patient or the legal guardian
6. Willingness and ability to comly with the treatment plan, follow-up and laboratory tests as required

Exclusion Criteria:

1. Congenital aplastic anemia
2. Pregnancy or breastfeeding
3. Participated in other clinical trials within three months
4. Presence of Any fatal disease, including respiratory failure, heart failure, liver or kidney failure, et al
5. Aplastic anemia caused by the treatment of other malignant tumor treatment
6. With severe mental illness
7. With other malignant tumor
8. Severe infection or the infection difficult to be controlled
9. Received ATG or cyclosporine A within six months
10. Severely allergic to biological agents
11. Any other situation judged by the investigator that the patients inappropriate for entry into this study

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
The total response rate | Every 3 months to 24 months
  Response rate is the ratio of CR and PR patients to all evaluated patients at the time point. CR,PR,NR and relapse is evaluated according to the guidelines for the diagnosis and management of adult aplastic anaemia from British Committee for Standards in Haematology (BCSH)

SECONDARY OUTCOMES:
Neutrophil recovery time | From day 0 until the ﬁrst of 3 consecutive days
  The neutrophil recovery day is defined from day "0" until the ﬁrst of 3 consecutive days during which the absolute neutrophil count (ANC) is >0.5×10^9/L, without G-CSF administration .
Infection rates | 1 year
Overall survival | 2 years
Treatment related mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fang Zhou, MD, Study Chair — The General Hospital Of Jinan Military Command
Locations (1):
- The General Hospital Of Jinan Military Command, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Killick SB, Bown N, Cavenagh J, Dokal I, Foukaneli T, Hill A, Hillmen P, Ireland R, Kulasekararaj A, Mufti G, Snowden JA, Samarasinghe S, Wood A, Marsh JC; British Society for Standards in Haematology. Guidelines for the diagnosis and management of adult aplastic anaemia. Br J Haematol. 2016 Jan;172(2):187-207. doi: 10.1111/bjh.13853. Epub 2015 Nov 16. No abstract available. PMID 26568159
- [Result] Zhou F, Ge L, Yu Z, Fang Y, Kong F. Clinical observations on intensive immunosuppressive therapy combined with umbilical cord blood support for the treatment of severe aplastic anemia. J Hematol Oncol. 2011 Jun 10;4:27. doi: 10.1186/1756-8722-4-27. PMID 21663651
- [Result] Xie LN, Fang Y, Yu Z, Song NX, Kong FS, Liu XM, Zhou F. Increased immunosuppressive treatment combined with unrelated umbilical cord blood infusion in children with severe aplastic anemia. Cell Immunol. 2014 May-Jun;289(1-2):150-4. doi: 10.1016/j.cellimm.2014.03.014. Epub 2014 Apr 3. PMID 24838091
- [Result] Yu Z, Zhou F, Ge LF, Liu XM, Fang Y, Xie LN, Kong FS, Song NX, Yu QQ. Mechanism of immunosuppressants combined with cord blood for severe aplastic anemia. Int J Clin Exp Med. 2015 Feb 15;8(2):2484-94. eCollection 2015. PMID 25932194
- [Result] Xie LN, Zhou F. Unexpected unrelated umbilical cord blood stem cell engraft in two patients with severe aplastic anemia that received immunosuppressive treatment: A case report and literature review. Exp Ther Med. 2015 Oct;10(4):1563-1565. doi: 10.3892/etm.2015.2698. Epub 2015 Aug 21. PMID 26622526